CLINICAL TRIAL: NCT03943095
Title: Randomized Controlled Examiner-Blind Phase II Exploratory Clinical Study to Characterize the Efficacy Profile of an Experimental Dual Active Combination Dentifrice for the Relief of Dentin Hypersensitivity, in Subjects With Clinically Diagnosed Dentin Hypersensitivity
Brief Title: Study to Characterize the Efficacy of a Dual Active Dentifrice for the Relief of Dentin Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 209723; 209723 (Other: GlaxoSmithKline)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Dentin Hypersensitivity; Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate; Tin Fluorides

STUDY DESIGN:
Intervention Model Description: Single center, 8-week, randomized, controlled, parallel design, exploratory clinical study in healthy participants with dentin hypersensitivity. Eligible participants will be stratified by the maximum Baseline Schiff sensitivity score of their two selected test teeth).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examiner-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Dentifrice (Experimental): Participants will be instructed to apply a strip of dentifrice (a full brush head) containing 5 % weight by weight (w/w) potassium nitrate and 0.454% w/w stannous fluoride (1100 parts per million [ppm] fluoride). Participants will brush their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and will be permitted to rinse with water post-brushing.
  Interventions: Other: Potassium Nitrate; Other: Stannous Fluoride
- Control Dentifrice (Active Comparator): Participants will be instructed to apply a strip of dentifrice (a full brush head) containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants will brush their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and will be permitted to rinse with water post-brushing.
  Interventions: Other: Stannous Fluoride

INTERVENTIONS:
Other: Potassium Nitrate — The test dentifrice contains 5% w/w potassium nitrate.
  Arms: Test Dentifrice
Other: Stannous Fluoride — The test and control dentifrices contain 0.454% w/w stannous fluoride (1100 ppm fluoride).

SUMMARY:
This exploratory study will characterize the efficacy profile of an experimental dual active 5 percent (%) potassium nitrate/0.454% stannous fluoride dentifrice, compared to a single active 0.454% stannous fluoride desensitizing dentifrice, over an 8-week treatment period.

DETAILED DESCRIPTION:
This will be a single center, 8-week, randomized, controlled, examiner-blind, two treatment arm, parallel design, stratified (by maximum Baseline Schiff sensitivity score of the two selected test teeth), Phase II, exploratory clinical study in healthy participants with DH. It is hypothesized that the combination of two antisensitivity active ingredients with complementary modes of action (potassium nitrate: nerve desensitization; stannous fluoride: dentin tubule occlusion) will deliver superior anti-sensitivity efficacy, compared to either active alone.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed
* Participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures
* Participant in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history, or upon oral examination, or condition that would impact the Participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements
* Male participant able to father children or female participant of child-bearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 5 days after the last dose of assigned treatment
* AT VISIT 1 (Screening): Participant must have

  1. a self-reported history of dentin hypersensitivity (DH) lasting more than six months but not more than 10 years
  2. a minimum of 20 natural teeth
  3. a minimum of 2 accessible, non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically diagnosed DH; each tooth must meet the following criteria:
* exposed dentin due to facial/cervical erosion, abrasion or gingival recession (EAR)
* Modified Gingival Index (MGI) score = 0 adjacent to the test area (exposed dentin) only
* Clinical mobility less than or equal to (=<) 1
* DH, as evidenced by qualifying levels of tactile and evaporative air sensitivity (tactile threshold [=<] 20 gram (g); Schiff sensitivity score greater than or equal to [>=] 2)
* AT VISIT 2 (Baseline):

Participant must have a minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), preferably in different quadrants, with DH, as evidenced by qualifying tactile and evaporative air sensitivity (each tooth must have a tactile threshold (=<) 20 g and a Schiff sensitivity score (>=) 2) at the Screening and Baseline visits

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a GlaxoSmithKline Consumer Healthcare (GSK CH) employee directly involved in the conduct of the study or a member of their immediate family
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical, oral, psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study
* Participant with any condition which, in the opinion of the investigator or medically qualified designee, causes xerostomia
* Participant who is a pregnant female (as evidenced by a positive Urine Pregnancy Test [UPT] at Screening)
* Participant who is a breast-feeding female
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participant with a recent history (within the last year) of alcohol or other substance abuse
* Participant who has participated in another tooth desensitizing treatment study within 8 weeks Screening
* Participant who has used an oral care product indicated for the relief of DH within 8 weeks of Screening (participant will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients)
* Participant who has had dental prophylaxis within 4 weeks of Screening
* Participant who has had a tooth bleaching procedure within 8 weeks of Screening
* Participant who has had treatment for periodontal disease (including surgery) within 12 months of Screening
* Participant who has had scaling or root planning within 3 months of Screening
* Participant with gross periodontal disease
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy
* Participant with a tongue or lip piercing or presence of multiple dental implants
* Participant with fixed or removable partial dentures
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer
* SPECIFIC DENTITION EXCLUSIONS FOR 'TEST TEETH':

  1. Tooth with evidence of current or recent caries or reported treatment of decay within 12 months of Screening
  2. Tooth with exposed dentin but with deep, defective or facial restorations
  3. Tooth with full crown or veneer
  4. Sensitive tooth with contributing etiologies other than erosion, abrasion or recession to exposed dentin
  5. Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Participant taking daily doses of medication/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with the perception of pain (examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs)
* AT VISIT 1 (Screening):

Participant who has taken antibiotics in the 2 weeks prior to the Screening visit

- AT VISIT 2 (Baseline): Participant who has taken antibiotics in the 2 weeks prior to the Baseline visit, during the acclimatization period

* Participant taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia
* Participant who requires antibiotic prophylaxis for dental procedures
* Participant who has previously been enrolled in this study
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Mississauga, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Canada
Pre-assignment Details: A total of 123 participates were screened and enrolled, out of which 104 participants were randomized in the study and 19 participants were not randomized.
Groups:
- Test Dentifrice: Participants were instructed to apply a strip of dentifrice (a full brush head) containing 5 percent (%) weight by weight (w/w) potassium nitrate and 0.454% w/w stannous fluoride (1100 parts per million [ppm] fluoride). Participants brushed their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and were permitted to rinse with water post-brushing.Participants received test dentifrice via a manual toothbrush throughout the study duration (8 weeks i.e. till Day 56) twice daily.
- Control Dentifrice: Participants were instructed to apply a strip of dentifrice (a full brush head) containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants brushed their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and were permitted to rinse with water post-brushing. Participants received control dentifrice via a manual toothbrush throughout the study duration (8 weeks i.e. till Day 56) twice daily.
Period: Overall Study
Arm/Group | Test Dentifrice | Control Dentifrice
Started | 52 | 52
Completed | 51 | 51
Not Completed | 1 | 1
Not completed — Incorrectly dispensed wrong box kit | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all randomized participants who received at least one dose of study product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice | Control Dentifrice | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (10.70) | 51.3 (10.45) | 51.3 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 50 | 52 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 21 | 36
  White | 31 | 26 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Baseline (Day 0)
Description: Evaporative air sensitivity was assessed on facial surfaces of eligible incisor,canine and pre-molar teeth by directing a one second application of air from standard dental syringe held perpendicular to tooth surface, approximately 1-2 millimeter (mm) coronal to the gingival margin from a distance of approximately 1 centimeter (cm).Participant response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative air stimulus.0=Does not respond to air stimulation;1=Responds to air stimulus but does not request discontinuation of stimulus;2=Responds to air stimulus and requests discontinuation or moves from stimulus;3=Responds to stimulus,considers stimulus to be painful, requests discontinuation of the stimulus. Score range 0-3; a decrease in Schiff sensitivity score indicates an improvement.Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Baseline (Day 0)
Population: A modified Intent-to-Treat (mITT) population included all randomized participants who received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Test Dentifrice: Participants were instructed to apply a strip of dentifrice (a full brush head) containing 5 percent (%) weight by weight (w/w) potassium nitrate and 0.454% w/w stannous fluoride (1100 parts per million [ppm] fluoride). Participants brushed their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and were permitted to rinse with water post-brushing.
- Control Dentifrice: Participants were instructed to apply a strip of dentifrice (a full brush head) containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants brushed their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and were permitted to rinse with water post-brushing.
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 2.61 (0.063) | 2.60 (0.063)

2. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 3
Description: Evaporative air sensitivity was assessed on facial surfaces of eligible incisor,canine and pre-molar teeth by directing a one second application of air from a standard dental syringe held perpendicular to the tooth surface, approximately 1-2 mm coronal to the gingival margin, and from a distance of approximately 1 cm. Participant response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative air stimulus. 0=Does not respond to air stimulation;1=Responds to air stimulus but does not request discontinuation of stimulus;2=Responds to air stimulus and requests discontinuation or moves from stimulus;3=Responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Score range 0-3; a decrease in Schiff sensitivity score indicates an improvement. Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Day 3
Population: mITT population included all randomized participants who received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Test Dentifrice: Participants were instructed to apply a strip of dentifrice (a full brush head) containing 5 % w/w potassium nitrate and 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants brushed their two selected 'test teeth' first, followed by the whole mouth for at least one timed minute, twice daily (morning and evening), and were permitted to rinse with water post-brushing.
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 1.19 (0.104) | 1.46 (0.104)

3. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 7
Description: as for outcome 2
Time Frame: Day 7
Population: mITT population included all randomized participants who received at least one dose of study product and had at least one post-baseline efficacy measurement.Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 0.73 (0.097) | 1.20 (0.120)

4. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 14
Description: as for outcome 2
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 0.52 (0.085) | 1.07 (0.134)

5. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 28
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 0.32 (0.087) | 0.75 (0.121)

6. Primary Outcome: Mean Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Day 56
Description: as for outcome 2
Time Frame: Day 56
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | 0.12 (0.043) | 0.42 (0.100)

7. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Baseline (Day 0)
Description: Tactile sensitivity was assessed for eligible incisor,canine and pre-molar teeth using a constant pressure probe (Yeaple probe),starting at 10 gram (g) and rising in increments of 10 g until the tactile threshold or maximum force for that visit is reached.The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine.After each application,the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response).The pressure setting at which participant gave two consecutive 'yes' responses was recorded as the tactile threshold (g).At Baseline, the maximum force was 20 g;at all subsequent visits, 80 g.If no sensitivity was found at the upper limit,the tactile threshold is recorded as greater than (>) 20 g (baseline) or >80 g (all other visits).An increase in tactile threshold indicates an improvement.Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Baseline (Day 0)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 11.06 (0.372) | 12.31 (0.574)

8. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 3
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe),starting at 10 g and rising in increments of 10 g until the tactile threshold or maximum force for that visit is reached. The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine.After each application, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline,the maximum force is 20 g; at all subsequent visits, 80 g. If no sensitivity was found at the upper limit,the tactile threshold is recorded as greater than (>) 20 g (baseline) or >80 g (all other visits). An increase in tactile threshold indicates an improvement.Mean was calculated once by selecting two test teeth which were located in different quadrants of mouth.
Time Frame: Day 3
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 31.35 (2.087) | 27.98 (2.061)

9. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 7
Description: as for outcome 8
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 47.45 (3.075) | 38.75 (2.983)

10. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 14
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 60.59 (3.271) | 48.53 (3.549)

11. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 28
Description: as for outcome 8
Time Frame: Day 28
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 71.67 (3.044) | 57.94 (4.076)

12. Primary Outcome: Mean Tactile Threshold (Average of the Two Selected Test Teeth) at Day 56
Description: as for outcome 8
Time Frame: Day 56
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 79.71 (2.390) | 64.80 (3.921)

13. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score Greater Than or Equal to [>=] 1) on Day 0 (Baseline)
Description: Number of eligible teeth were identified at screening with Schiff sensitivity score of >=1 (Schiff sensitivity scale: 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3=Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus). A decrease in the number of sensitive teeth indicates an improvement.
Time Frame: Baseline (Day 0)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of sensitive teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of sensitive teeth | 3.1 (0.14) | 3.2 (0.15)

14. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 3
Description: as for outcome 13
Time Frame: Day 3
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of Sensitive Teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of Sensitive Teeth | 3.6 (0.20) | 3.6 (0.22)

15. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 7
Description: as for outcome 13
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Number of Sensitive teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of Sensitive teeth | 2.2 (0.26) | 3.2 (0.26)

16. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 14
Description: as for outcome 13
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Number of Sensitive teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of Sensitive teeth | 1.7 (0.24) | 2.8 (0.29)

17. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 28
Description: as for outcome 13
Time Frame: Day 28
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Number of Sensitive teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of Sensitive teeth | 1.0 (0.23) | 2.1 (0.30)

18. Primary Outcome: Number of Sensitive Teeth (Schiff Sensitivity Score >= 1) on Day 56
Description: as for outcome 13
Time Frame: Day 56
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Number of Sensitive teeth
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Number of Sensitive teeth | 0.5 (0.15) | 1.3 (0.25)

19. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Day 56
Description: Evaporative air sensitivity was assessed on the facial surfaces of teeth by directing one second application of air from dental syringe held perpendicular to tooth surface, approximately 1-2 mm coronal to gingival margin and from a distance of approximately 1 cm. Participant response to stimulus was evaluated using Schiff sensitivity scale following administration of the evaporative air stimulus.0=Does not respond to air stimulation;1=Responds to air stimulus but does not request discontinuation of stimulus;2=Responds to air stimulus and requests discontinuation or moves from stimulus;3=Responds to stimulus, considers stimulus to be painful, requests discontinuation of stimulus. Score range 0-3;a decrease in Schiff sensitivity score indicates improvement. Adjusted mean change from baseline are derived from analysis of covariance (ANCOVA) model which included treatment as a factor and baseline Schiff sensitivity score as a covariate with change from baseline as dependent variable.
Time Frame: Baseline (Day 0), Day 56
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Score on a scale | -2.48 (0.073) | -2.17 (0.073)

20. Secondary Outcome: Change From Baseline (Day 0) in Tactile Threshold on Day 56
Description: Tactile sensitivity was assessed for eligible teeth using constant pressure probe (Yeaple probe),starting at 10 g and rising in increments of 10 g until tactile threshold for that visit is reached. The probe tip was placed perpendicular to facial surface of tooth and drawn slowly across exposed dentine. After each application, participant was asked whether they experienced any pain or discomfort (yes/no response).The pressure setting at which participant gives two consecutive 'yes' responses was recorded as the tactile threshold (g).At Baseline, the maximum force was 20g;at all subsequent visits,80g.If no sensitivity was found at the upper limit, the tactile threshold was recorded as >20 g (Baseline) or >80 g (all other visits).An increase in tactile threshold indicates an improvement. Adjusted mean change from baseline are derived from ANCOVA model which included treatment as factor and baseline tactile senstivity as covariate with change from baseline as dependent variable.
Time Frame: Baseline (Day 0), Day 56
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 52 | 52
Grams | 69.34 (3.067) | 51.94 (3.067)

ADVERSE EVENTS:
Time Frame: From screening up to Day 56
Description: Safety population: all participants who were eligible to participate in the study and received at least one dose of study medication. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported. A participant with multiple occurrences of AEs counted once in AE category. A participant with multiple AEs within a primary system organ class was counted once in system organ class.
Arm/Group | Test Dentifrice | Control Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 2/52 | 1/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Dentifrice (N=52) | Control Dentifrice (N=52)
Oral mucosal exfoliation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03943095/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03943095/SAP_001.pdf